CLINICAL TRIAL: NCT06204224
Title: Personal Variables Affecting the Successful Aging Level of Individuals Age of Sixty and Over
Brief Title: Personal Variables Affecting the Successful Aging
Status: Completed | Type: Observational
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğu Usanma Koban, asst. prof., Marmara University Pendik Training and Research Hospital
Other Study IDs: 2018/107
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Aging; Healthy Lifestyle; Coping Skills
Keywords: successful aging; aging; healthy aging; family medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Three hundreds patients aged 60 years and older applicant for any reasons between January 3, 2019 and May 30, 2019, in Health Sciences University Haydarpaşa Numune Training and Research Hospital Family Medicine Polyclinics. A 21-item questionnaire including demographic information was asked to the individuals who gave consent to participate in the study, voluntarily, and who met the participation criteria and the Successful Aging Scale was administered face-to-face with the questionnaire method. Participants were evaluated under two subheadings according to the Successful Aging Scale and the results were compared with their demographic characteristics.

DETAILED DESCRIPTION:
In our cross-sectional study; the target sample size was calculated as 299, with a population of 1350. The prevalence was 50%, the standard error was 5% in a 95% confidence interval. Between 03.01.2019 and 30.05.2019; 300 elderly volunteers who applied to the Health Sciences University Haydarpaşa Numune Training and Research Hospital Family Medicine Polyclinics for any reason, who were not diagnosed with neuropsychiatric disease, do not had physical or mental problems that would prevent them from understanding and filling the scales and do not have a health problem that require urgent intervention are included. Participants were informed, their consent was taken, and a 21-item sociodemographic form prepared by the researchers was applied. Afterwards, a 7-point Likert-type "Successful Aging Scale" (SAS) consisting of 10 questions was applied to the participants.16 The scale had two sub-components, namely "healthy lifestyle" (HL) and "adaptive coping" (AC). The values of the expressions in the scale were as "strongly agree:7, agree:6, partially agree:5, undecided:4, partially disagree:3, disagree:2, strongly disagree:1". The values for each individual were summed up and the scale was evaluated by subtracting the total score. Finally, the results from the questionnaire and the Successful Aging Scale were compared and analyzed according to subcomponents.

ELIGIBILITY:
Inclusion Criteria:

* Not having received a diagnosis of dementia at any stage of life.
* Not having any cognitive or physical impediments that hinder understanding and completing the scales.
* Having full orientation and cooperation.
* Having completed the scales in their entirety.
* The absence of symptoms or diseases requiring urgent intervention.
* Voluntarily participating in the study and having signed the informed consent form after being informed.

Exclusion Criteria:

* Having received a diagnosis of dementia.
* Having cognitive and physical impediments that hinder understanding the scales.
* Lack of full orientation and cooperation.
* Having a clinically significant diagnosis of an active psychiatric disorder.
* having symptoms of a situation requiring urgent intervention.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 60 and above, who presented to the Family Medicine Clinics of Haydarpaşa Numune Training and Research Hospital between January 3, 2019, and May 30, 2019, for any reason; and voluntarily agreed to participate, were included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Sociodemographic properties affect successful aging scores | 1 week
  Gender, education level, level of income, retirement status affect scores of "Successful Aging Scale" (SAS) was used to assess the participants. The SAS consisted of 10 questions and had two sub-components: "healthy lifestyle" (HL) and "adaptive coping" (AC). The scale utilized the following response options: "strongly agree" (7), "agree" (6), "partially agree" (5), "undecided" (4), "partially disagree" (3), "disagree" (2), and "strongly disagree" (1). The higher the score taken from the scale, the higher the level of successful aging.

SECONDARY OUTCOMES:
Healthy life habits affect successful aging scores | 1 week
  Doing sports regularly, quitting existing bad habits (smoking and alcohol consumption) affect scores of "Successful Aging Scale" (SAS) was used to assess the participants. The SAS consisted of 10 questions and had two sub-components: "healthy lifestyle" (HL) and "adaptive coping" (AC). The scale utilized the following response options: "strongly agree" (7), "agree" (6), "partially agree" (5), "undecided" (4), "partially disagree" (3), "disagree" (2), and "strongly disagree" (1). The higher the score taken from the scale, the higher the level of successful aging.
Having chronic diseases affect successful aging scores | 1 week
  Having hypertension, diabetes, cardiovascular disease, hyperlipidemia, chronic obstructive pulmonary disease (COPD), kidney failure, thyroid diseases and other chronic diseases affect scores of "Successful Aging Scale" (SAS) was used to assess the participants. The SAS consisted of 10 questions and had two sub-components: "healthy lifestyle" (HL) and "adaptive coping" (AC). The scale utilized the following response options: "strongly agree" (7), "agree" (6), "partially agree" (5), "undecided" (4), "partially disagree" (3), "disagree" (2), and "strongly disagree" (1). The higher the score taken from the scale, the higher the level of successful aging.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Research and Training Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McLaughlin SJ, Jette AM, Connell CM. An examination of healthy aging across a conceptual continuum: prevalence estimates, demographic patterns, and validity. J Gerontol A Biol Sci Med Sci. 2012 Jun;67(7):783-9. doi: 10.1093/gerona/glr234. Epub 2012 Feb 24. PMID 22367432
- [Background] Iwamasa GY, Iwasaki M. A new multidimensional model of successful aging: perceptions of Japanese American older adults. J Cross Cult Gerontol. 2011 Sep;26(3):261-78. doi: 10.1007/s10823-011-9147-9. PMID 21626301
- [Background] Park SM, Jang SN, Kim DH. Gender differences as factors in successful ageing: a focus on socioeconomic status. J Biosoc Sci. 2010 Jan;42(1):99-111. doi: 10.1017/S0021932009990204. Epub 2009 Aug 25. PMID 19703332
- [Background] Cosco TD, Stephan BCM, Brayne C, Muniz G; MRC CFAS. Education and Successful Aging Trajectories: A Longitudinal Population-Based Latent Variable Modelling Analysis. Can J Aging. 2017 Dec;36(4):427-434. doi: 10.1017/S0714980817000344. Epub 2017 Oct 11. PMID 29019302